CLINICAL TRIAL: NCT05781412
Title: Modulation of the Activity in the Cerebellum With Transcranial Direct Current Stimulation in Autistic Participants
Brief Title: Modulation of the Activity of the Cerebellum in Autism (MACA)
Acronym: MACA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beatriz Catoira (Other)
Collaborators: Vrije Universiteit Brussel (Other); University Ghent (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor-Investigator, Beatriz Catoira, MsC, PhD student at the Vrije Universiteit Brussel, Vrije Universiteit Brussel
Organization: Vrije Universiteit Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22064MACA
Record Dates: First submitted 2022-12-06; First posted 2023-03-23 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder
Keywords: tDCS; Cerebellum; neuromodulation; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: There will be three groups of participants: autism-diagnosed, autism-non-diagnosed and neurotypical individuals (healthy controls). On each group, participants will be randomly allocated to one of two groups: anodal stimulation in the first session or anodal stimulation in the second session (in the other session there will be sham stimulation).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ASD_anodalstimulation (Active Comparator): ASD participant, anodal stimulation on the first session, sham stimulation on the second sesion
  Interventions: Device: tDCS
- ASD_shamstimulation (Sham Comparator): ASD participant, sham stimulation on the first session, anodal stimulation on the second sesion
  Interventions: Device: tDCS
- NT_anodalstimulation (Active Comparator): Neurotypical participant, anodal stimulation on the first session, sham stimulation on the second sesion
  Interventions: Device: tDCS
- NT_shamstimulation (Sham Comparator): Neurotypical participant, sham stimulation on the first session, anodal stimulation on the second sesion
  Interventions: Device: tDCS
- H-AQ_anodalstimulation (Active Comparator): non diagnosed autistic participant,anodal stimulation on the first session, sham stimulation on the second sesion
  Interventions: Device: tDCS
- H-AQ_shamstimulation (Sham Comparator): non diagnosed autistic participant, sham stimulation on the first session, anodal stimulation on the second sesion
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Anodal and Sham cerebellar tDCS will be used in each participant in a counterbalanced order

SUMMARY:
Research on the involvement of the cerebellum in social understanding behavior and the mentalizing brain system has just begun. Knowledge about the neurobiology of social understanding is important for understanding the ways to manipulate these processes. Like cerebral tDCS, cerebellar tDCS could then be used to enhance more complex processes, such as mentalizing, in healthy individuals. It can eventually also be examined as a therapeutic tool for patients with mentalizing difficulties such as patients with ASD. In this study, it is examined whether anodal tDCS at the right posterior cerebellum influences social understanding and which cerebro-cerebellar networks play a role in this process.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are a group of lifelong neurodevelopmental disorders characterized by social and communicative difficulties and repetitive and stereotyped behaviors. Research has shown that cerebellar abnormalities are among the most important etiological factors for ASD. The cerebellum is found to be most frequently involved in tasks where participants must remember or imagine past or future autobiographical events, judge persons or situations based on behavioral sentences, make trait inferences of others using stories, words or faces, and describe persons or objects based on behavioral or object pictures. Recent research has also provided evidence on the involvement of the posterior areas of the cerebellum in social cognition.

Specifically, the areas crus I and crus II, located at the lateral hemispheres of the posterior cerebellum, are associated with more complex cognitive and social processes, such as mentalizing. Mentalizing is the cognitive ability to attribute mental states, such as desires, intentions, and beliefs, to other people. This ability is needed to understand and predict other people's behavior and is the main component of social cognition. Problems with mentalizing, including the attribution of false beliefs to others, are characteristic for autism spectrum disorder (ASD). A sequencing task (that included social and non social conditions) showing that cerebellar patients performed worse than healthy participants.

Facial emotion recognition refers to the ability to derive emotional meaning from facial expressions and has been shown to underlie social competency. Recent literature reviews have reported significant facial emotion recognition impairments in individuals with ASD. These impairments take various forms, such as a reduced accuracy in labeling facial emotions or reduced specificity in rating facial emotions of varying intensity . Thus, there is evidence suggesting that ASD is associated with a selective impairment in facial emotion recognition.

Transcranial direct current stimulation (tDCS) is a noninvasive technique that can produce long-lasting changes in the excitability and spontaneous activity of the stimulated brain areas. Therefore, tDCS is investigated as a possible treatment for different psychiatric diseases. Cerebellar tDCS have shown to also produce prolonged changes successfully at the neural and behavioral level. However, due to the high density of neurons in the cerebellum and diffuse connections to the cerebrum, it is more difficult to understand the working mechanisms of cerebellar as compared to cerebral tDCS. In addition, the electrical current will spread across more neurons in the cerebellum by cerebellar tDCS and will functionally affect the cerebral regions to which these cerebellar neurons are connected as well. Therefore, the type of behavioral effect, such as an improvement of performance after anodal tDCS or an impairment of performance after cathodal tDCS, is harder to predict for cerebellar than cerebral tDCS.

Modulation of social understanding with tDCS has been studied by stimulating the key mentalizing regions mPFC and TPJ. In healthy participants, an improvement on tasks was found that required the enhancement or inhibition of representation of the self or of others, which is important for mentalizing, after anodal tDCS at the TPJ compared to sham tDCS or cathodal tDCS. The effect of cerebellar tDCS on social understanding using action sequences has not yet been examined.

ELIGIBILITY:
Participant Inclusion/exclusion criteria:

* Participants must be more than 18 years old
* normal eyesight and hearing;
* Dutch, French or English speaking;

Neurotypical participants inclusion/exclusion criteria:

* No disorder (now or in the past) that could have affected the brain such as cerebrovascular accidents (CVA), neurodegenerative disorders, or essential tremor;
* No neurological diseases that could affect reasoning or intellectual abilities (such as Parkinson's Disease, Epilepsy, and Multiple Sclerosis)
* Neurotypical participants will be matched on age and gender to the ASD population;

ASD participants inclusion/exclusion criteria:

Patients with a formal diagnosis of high-functioning ASD as determined by the clinical psychologist/psychiatrist.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
PS_RT | assessment will begin 10 minutes after stimulation and last up to 15 minutes
  Reaction Time in the pictorial sequencing time
PS_accuracy | assessment will begin 10 minutes after stimulation and last up to 15 minutes
  Accuracy in the pictorial sequencing task
ER_RT | assessment will begin 20 minutes after stimulation and last up to 5 minutes
  Reaction Times in the emotion recognition task
ER_accuracy | assessment will begin 20 minutes after stimulation and last up to 5 minutes
  Accuracy in the emotion recognition task
Brain activity at the emotion recognition task | assessment will begin 20 minutes after stimulation and last up to 5 minutes
  Brain activity (fMRI) in regions of interest/whole brain analysis. Differences between stimulation and sham, between task conditions and between sessions as well as possible interactions in between those factors and covariates (AQ scores, age, gender...)
Brain activity at resting state | assesment will begin concurrent with stimulation and last up to 20 minutes
  Brain activity (fMRI) in regions of interest/whole brain analysis. Differences between stimulation and sham, between task conditions and between sessions as well as possible interactions in between those factors and covariates (AQ scores, age, gender...)
Brain activity at the pictorial sequencing task | assessment will begin 10 minutes after stimulation and last up to 15 minutes
  Brain activity (fMRI) in regions of interest/whole brain analysis. Differences between stimulation and sham, between task conditions and between sessions as well as possible interactions in between those factors and covariates (AQ scores, age, gender...)
White matter integrity in the cerebellum | assessment will begin immediately after stimulation and last up to 10 minutes
  White matter integrity matrix (FA, MD, RD) in the cerebellum using tract-based spatial statistics in the cerebellum & differences between groups

SECONDARY OUTCOMES:
Connectivity_PStask | assessment will begin 10 minutes after stimulation and last up to 15 minutes
  Brain connectivity (fMRI) analysis on the pictorial sequencing task
Connectivity_ERtask | assessment will begin 20 minutes after stimulation and last up to 5 minutes
  Brain connectivity (fMRI) analysis on the emotion recognition task
Connectivity_stimulation | assesment will begin concurrent with stimulation and last up to 20 minutes
  Brain connectivity (fMRI) analysis during stimulation
Fiber tractography between the cerebellum and the default mode/ mentalizing network | assessment will begin immediately after stimulation and last up to 10 minutes
  Fiber tractography (Diffusion weighted imaging) between the cerebellum and the default mode / mentalizing network, by extraction of white matter integrity parameters on each fiber tract
ROI-based structural connectivity | assessment will begin immediately after stimulation and last up to 10 minutes
  Structural connectivity (DWI) between ROIs from the default mode/mentalizing network
Whole brain structural network construction | assessment will begin immediately after stimulation and last up to 10 minutes
  Structural connectivity (DWI) within the whole brain using graph theory

OTHER OUTCOMES:
Electrical Field Simulations | First 10 minutes of assessment
  Simulation of the electric field generated by the tDCS stimulation.
Correlations between DWI, behavioural data, simulation and functional data | assessment will include data from the 60 minutes that are spent in the scanner in the session
  The primary outcome measures from the diffusion weighted imaging will provide different measures for structural connectivity per participant. The correlation of these measures with behavioural and/or functional data will be computed.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Van Overwalle F, Baetens K, Marien P, Vandekerckhove M. Social cognition and the cerebellum: a meta-analysis of over 350 fMRI studies. Neuroimage. 2014 Feb 1;86:554-72. doi: 10.1016/j.neuroimage.2013.09.033. Epub 2013 Sep 27. PMID 24076206
- [Result] Buckner RL, Krienen FM, Castellanos A, Diaz JC, Yeo BT. The organization of the human cerebellum estimated by intrinsic functional connectivity. J Neurophysiol. 2011 Nov;106(5):2322-45. doi: 10.1152/jn.00339.2011. Epub 2011 Jul 27. PMID 21795627
- [Result] Murphy CM, Wilson CE, Robertson DM, Ecker C, Daly EM, Hammond N, Galanopoulos A, Dud I, Murphy DG, McAlonan GM. Autism spectrum disorder in adults: diagnosis, management, and health services development. Neuropsychiatr Dis Treat. 2016 Jul 7;12:1669-86. doi: 10.2147/NDT.S65455. eCollection 2016. PMID 27462160
- [Result] Murphy DG, Beecham J, Craig M, Ecker C. Autism in adults. New biologicial findings and their translational implications to the cost of clinical services. Brain Res. 2011 Mar 22;1380:22-33. doi: 10.1016/j.brainres.2010.10.042. Epub 2010 Oct 20. PMID 20969835
- [Result] D'Mello AM, Stoodley CJ. Cerebro-cerebellar circuits in autism spectrum disorder. Front Neurosci. 2015 Nov 5;9:408. doi: 10.3389/fnins.2015.00408. eCollection 2015. PMID 26594140
- [Result] Fatemi SH, Aldinger KA, Ashwood P, Bauman ML, Blaha CD, Blatt GJ, Chauhan A, Chauhan V, Dager SR, Dickson PE, Estes AM, Goldowitz D, Heck DH, Kemper TL, King BH, Martin LA, Millen KJ, Mittleman G, Mosconi MW, Persico AM, Sweeney JA, Webb SJ, Welsh JP. Consensus paper: pathological role of the cerebellum in autism. Cerebellum. 2012 Sep;11(3):777-807. doi: 10.1007/s12311-012-0355-9. PMID 22370873
- [Result] Sathyanesan A, Zhou J, Scafidi J, Heck DH, Sillitoe RV, Gallo V. Emerging connections between cerebellar development, behaviour and complex brain disorders. Nat Rev Neurosci. 2019 May;20(5):298-313. doi: 10.1038/s41583-019-0152-2. PMID 30923348
- [Result] Heleven E, van Dun K, Van Overwalle F. The posterior Cerebellum is involved in constructing Social Action Sequences: An fMRI Study. Sci Rep. 2019 Jul 31;9(1):11110. doi: 10.1038/s41598-019-46962-7. PMID 31366954
- [Result] Van Overwalle F, Van de Steen F, Marien P. Dynamic causal modeling of the effective connectivity between the cerebrum and cerebellum in social mentalizing across five studies. Cogn Affect Behav Neurosci. 2019 Feb;19(1):211-223. doi: 10.3758/s13415-018-00659-y. PMID 30361864
- [Result] Leggio M, Olivito G. Topography of the cerebellum in relation to social brain regions and emotions. Handb Clin Neurol. 2018;154:71-84. doi: 10.1016/B978-0-444-63956-1.00005-9. PMID 29903453
- [Result] Frith CD, Frith U. Interacting minds--a biological basis. Science. 1999 Nov 26;286(5445):1692-5. doi: 10.1126/science.286.5445.1692. PMID 10576727
- [Result] Mier D, Lis S, Neuthe K, Sauer C, Esslinger C, Gallhofer B, Kirsch P. The involvement of emotion recognition in affective theory of mind. Psychophysiology. 2010 Nov;47(6):1028-39. doi: 10.1111/j.1469-8986.2010.01031.x. PMID 20456660
- [Result] Baron-Cohen S, Leslie AM, Frith U. Does the autistic child have a "theory of mind"? Cognition. 1985 Oct;21(1):37-46. doi: 10.1016/0010-0277(85)90022-8. No abstract available. PMID 2934210
- [Result] Leggio MG, Tedesco AM, Chiricozzi FR, Clausi S, Orsini A, Molinari M. Cognitive sequencing impairment in patients with focal or atrophic cerebellar damage. Brain. 2008 May;131(Pt 5):1332-43. doi: 10.1093/brain/awn040. Epub 2008 Mar 11. PMID 18334535
- [Result] Izard C, Fine S, Schultz D, Mostow A, Ackerman B, Youngstrom E. Emotion knowledge as a predictor of social behavior and academic competence in children at risk. Psychol Sci. 2001 Jan;12(1):18-23. doi: 10.1111/1467-9280.00304. PMID 11294223
- [Result] Uljarevic M, Hamilton A. Recognition of emotions in autism: a formal meta-analysis. J Autism Dev Disord. 2013 Jul;43(7):1517-26. doi: 10.1007/s10803-012-1695-5. PMID 23114566
- [Result] Kennedy DP, Adolphs R. The social brain in psychiatric and neurological disorders. Trends Cogn Sci. 2012 Nov;16(11):559-72. doi: 10.1016/j.tics.2012.09.006. Epub 2012 Oct 6. PMID 23047070
- [Result] Morya E, Monte-Silva K, Bikson M, Esmaeilpour Z, Biazoli CE Jr, Fonseca A, Bocci T, Farzan F, Chatterjee R, Hausdorff JM, da Silva Machado DG, Brunoni AR, Mezger E, Moscaleski LA, Pegado R, Sato JR, Caetano MS, Sa KN, Tanaka C, Li LM, Baptista AF, Okano AH. Beyond the target area: an integrative view of tDCS-induced motor cortex modulation in patients and athletes. J Neuroeng Rehabil. 2019 Nov 15;16(1):141. doi: 10.1186/s12984-019-0581-1. PMID 31730494
- [Result] Ferrucci R, Priori A. Transcranial cerebellar direct current stimulation (tcDCS): motor control, cognition, learning and emotions. Neuroimage. 2014 Jan 15;85 Pt 3:918-23. doi: 10.1016/j.neuroimage.2013.04.122. Epub 2013 May 9. PMID 23664951
- [Result] O'Reilly JX, Beckmann CF, Tomassini V, Ramnani N, Johansen-Berg H. Distinct and overlapping functional zones in the cerebellum defined by resting state functional connectivity. Cereb Cortex. 2010 Apr;20(4):953-65. doi: 10.1093/cercor/bhp157. Epub 2009 Aug 14. PMID 19684249
- [Result] van Dun K, Bodranghien FC, Marien P, Manto MU. tDCS of the Cerebellum: Where Do We Stand in 2016? Technical Issues and Critical Review of the Literature. Front Hum Neurosci. 2016 May 11;10:199. doi: 10.3389/fnhum.2016.00199. eCollection 2016. PMID 27242469
- [Result] Oldrati V, Schutter DJLG. Targeting the Human Cerebellum with Transcranial Direct Current Stimulation to Modulate Behavior: a Meta-Analysis. Cerebellum. 2018 Apr;17(2):228-236. doi: 10.1007/s12311-017-0877-2. PMID 28786014
- [Result] Santiesteban I, Banissy MJ, Catmur C, Bird G. Enhancing social ability by stimulating right temporoparietal junction. Curr Biol. 2012 Dec 4;22(23):2274-7. doi: 10.1016/j.cub.2012.10.018. Epub 2012 Nov 1. PMID 23122848
- [Result] Hogeveen J, Obhi SS, Banissy MJ, Santiesteban I, Press C, Catmur C, Bird G. Task-dependent and distinct roles of the temporoparietal junction and inferior frontal cortex in the control of imitation. Soc Cogn Affect Neurosci. 2015 Jul;10(7):1003-9. doi: 10.1093/scan/nsu148. Epub 2014 Dec 5. PMID 25481003
- [Result] Rogers TD, McKimm E, Dickson PE, Goldowitz D, Blaha CD, Mittleman G. Is autism a disease of the cerebellum? An integration of clinical and pre-clinical research. Front Syst Neurosci. 2013 May 10;7:15. doi: 10.3389/fnsys.2013.00015. eCollection 2013. PMID 23717269
- [Result] Yeung MK, Lee TL, Chan AS. Impaired Recognition of Negative Facial Expressions is Partly Related to Facial Perception Deficits in Adolescents with High-Functioning Autism Spectrum Disorder. J Autism Dev Disord. 2020 May;50(5):1596-1606. doi: 10.1007/s10803-019-03915-3. PMID 30758693

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT05781412/Prot_ICF_000.pdf